CLINICAL TRIAL: NCT02579317
Title: Project IMPACT: In-the-Moment Protection From Automatic Capture by Trigger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jennifer Buckman, Principal Investigator, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-015R; 1R01AA023667-01 (NIH)
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Substance Use Disorder
Keywords: Baroreflex mechanism; Alcohol Use Disorder; Substance Use Disorder; Heart Rate Variability; Breathing
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resonance Breathing (Experimental): Breathing is paced to the cardiovascular resonance frequency where heart, respiratory, and brain signals become aligned. This can potentially positively impact cognitive-emotional functioning.
  Interventions: Behavioral: Resonance Breathing
- Non-Resonance Breathing (Placebo Comparator): Breathing is paced at a non-resonance frequency. It does not align heart, respiratory, and brain signals, and thus does not impact cognitive-emotional functioning.
  Interventions: Behavioral: Non-Resonance Breathing

INTERVENTIONS:
Behavioral: Resonance Breathing — Breathing is paced with a pre-installed iPhone app that includes a visual pacer.
  Arms: Resonance Breathing
Behavioral: Non-Resonance Breathing — Breathing is paced with a pre-installed iPhone app that includes a visual pacer.
  Arms: Non-Resonance Breathing

SUMMARY:
Despite conscious intentions to remain abstinent, persons with substance use disorders often find that negative emotions and environmental cues automatically "trigger" drinking and other substance use. This study aims to test whether activating the baroreflex mechanism can be used "in the moment" to help resist drinking triggers. It consists of 3 phases (Recruitment, Intervention, Follow-up).

Stage 1: Trained research staff conduct a comprehensive clinical interview and questionnaires to assess participant's mood, substance use, and triggers. Participants are paired with a Primary Research Clinician (PRC) who will work with them during the intervention.

Stage 2: Approximately 4 weeks after intake into the Center for Great Expectations Intensive Outpatient program, an 8-week intervention begins. Pre-and post-intervention laboratory sessions occur at Cardiac Neuroscience Laboratory, Center of Alcohol Studies, Piscataway, NJ. Some participants take part in pre- and post-intervention neuroimaging sessions (Rutgers University Brain Imaging Center, Newark, NJ). Participants are randomized into an active intervention or control group after the pre-intervention lab session. They are given an iPhone and trained to use a paced breathing app that is pre-loaded onto the phone. Participants in both groups use their app any time they anticipate or experience a trigger to drink or use drugs. Participants are compensated for their use of the app and the time for participation. To ensure that participants are correctly performing the paced breathing task, their PRC visit with them weekly to provide coaching sessions using a computer-based biofeedback program. During the 4th week, ECG and respiration data are collected. Participants also complete questionnaires about mood and triggers, and provide feedback on the usefulness of the app.

During the lab sessions, participants complete a series of questionnaires and ECG, blood pressure and respiration are collected during four 5-minute tasks (resting baseline, non-resonance breathing, resonance breathing, and visual processing/attention). During the neuroimaging sessions, participants are placed in the scanner for structural scans and four 5-minute tasks (as tasks as previously noted); ECG and blood pressure are recorded.

Stage 3: Participants are re-contacted 1 and 3 months after the intervention to complete questionnaires about their quality of life across multiple domains and the usefulness of the app.

ELIGIBILITY:
Inclusion Criteria:

* Women over age 18
* Women diagnosed with substance use disorder
* Women participating in IOP at Center for Great Expectations, New Brunswick, NJ

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-11; Primary Completion 2020-03 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Active Substance Use (self-report questionnaire) | Three Months

SECONDARY OUTCOMES:
Quality of Life (self-report questionnaire) | Three Months
  Social support, financial resources, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Buckman, Ph.D., Principal Investigator — Center of Alcohol Studies
Locations (1):
- Center of Alcohol Studies, Piscataway, New Jersey, United States

REFERENCES:
- [Derived] Price JL, Bates ME, Pawlak AP, Uhouse SG, Todaro SM, Morgano J, Buckman JF. Use and perceived usefulness of a just-in-time resonance breathing intervention adjunct for substance use disorder: Contextual and physiological predictors. Front Psychiatry. 2022 Sep 7;13:945751. doi: 10.3389/fpsyt.2022.945751. eCollection 2022. PMID 36159943

DOCUMENTS (1):
  • Informed Consent Form (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT02579317/ICF_000.pdf